CLINICAL TRIAL: NCT01258205
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 139 in Healthy Subjects and Subjects With Mild to Severe Crohn's Disease, and Pharmacodynamics of AMG 139 in Healthy Subjects and Subjects With Mild to Severe Crohn's Disease
Brief Title: Multiple Ascending Doses of AMG 139 in Healthy and Crohn's Disease Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20090519
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Crohn's Disease
Keywords: Amgen; AMG 139; Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — AMG 139

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part B (Experimental): One dose level of AMG 139 administered as a multiple doses IV in subjects with mild-severe Crohn's disease.
  Interventions: Drug: AMG 139
- Part A (Experimental): Three dose levels of AMG 139 administered as a multiple doses IV or SC in healthy subjects.
  Interventions: Drug: AMG 139

INTERVENTIONS:
Drug: AMG 139 — Four dose levels of AMG 139 administered as multiple doses IV or SC in healthy volunteers (Part A) and subjects with moderate-severe Crohn's disease (Part B).

SUMMARY:
The purpose of this study is to assess the safety and tolerability of AMG 139 following multiple intravenous (IV) or subcutaneous (SC) dose administration in healthy subjects and in subjects with mild to severe Crohn's disease (CD).

ELIGIBILITY:
Inclusion Criteria:

Part A - Healthy Subjects:

* Healthy male or female of non-reproductive potential subjects between 18 to 45 years-of-age
* Body mass index (BMI) between 18 and 32 kg/m2
* Normal or clinically acceptable physical examination, clinical laboratory values, and ECG
* Additional inclusion criteria apply

Part B - Crohn's Subjects:

* Male or female subjects with CD between 18 to 55 years-of-age
* Body mass index (BMI) between 18 and 32 kg/m2
* Normal or clinically acceptable physical examination (PE), clinical laboratory values, and ECG; clinically acceptable PE includes evidence of mild to severe CD
* Diagnosis of ileal or ileo-colonic CD for a minimum of 6 months
* Mild to severe CD defined by a Crohn's Disease Activity Index (CDAI) score equal to or greater than 180 and equal to or less than 450
* Elevated fecal calprotectin and CRP
* Additional inclusion criteria apply

Exclusion Criteria:

Parts A - Healthy Subjects:

* History or evidence of a clinically significant disorder (including psychiatric), condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion;
* Recent or on-going infection(s)
* Underlying condition(s) that predisposes the subject to infections
* History of malignancy of any type
* Additional exclusion criteria apply

Part B only - Crohn's Subjects:

* History or evidence of a clinically significant disorder (including psychiatric), condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion;
* Recent or on-going infection(s)
* Underlying condition(s) that predisposes the subject to infections
* History of malignancy of any type
* Additional exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-02-28 (Actual); Primary Completion 2015-02-18 (Actual); Study Completion 2015-02-18 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability: treatment-emergent AEs including clinically significant changes in physical examinations, safety lab tests, ECG, vital signs, or immunogenicity to AMG 139 | 36 weeks

SECONDARY OUTCOMES:
Characterization of the pharmacokinetic (PK) parameters (AUCtau, Cmax, tmax) for AMG 139 after multiple IV and SC dose administrations in healthy subjects and subjects with mild to severe CD | 36 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Stony Brook University Medical Center, Stony Brook, New York
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (3):
  - QPharm Pty Limited, Herston, Queensland
  - Clinical Medical and Analytical eXellence CMAX, Adelaide, South Australia
  - Centre for Clinical Studies (Alfred), Prahran, Victoria